CLINICAL TRIAL: NCT06121011
Title: A Global Prospective Observational Registry of Patients With Pompe Disease
Status: Recruiting | Type: Observational
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: POM-005
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — miglustat; GAA protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: US Export: No

GROUPS / COHORTS (3):
- Cipaglucosidase alfa/Miglustat-treated patients
  Interventions: Biological: Cipaglucosidase alfa; Drug: Miglustat
- Other Enyzme Replacement Therapy (ERT)-treated patients
  Interventions: Biological: Alglucosidase alfa or Avalglucosidase alfa
- Untreated patients (those who are not currently receiving any medical therapy for Pompe disease)
  Interventions: Other: Untreated

INTERVENTIONS:
Biological: Cipaglucosidase alfa — Enzyme Replacement Therapy (ERT) via intravenous infusion
  Other Names: ATB200, Pombiliti
  Groups: Cipaglucosidase alfa/Miglustat-treated patients
Drug: Miglustat — Participants received ATB200 co-administered with AT2221 (Miglustat)
  Other Names: AT2221, Opfolda
  Groups: Cipaglucosidase alfa/Miglustat-treated patients
Biological: Alglucosidase alfa or Avalglucosidase alfa — Patients prescribed other commercially available ERT after local regulatory approval
  Other Names: Myozyme, Lumizyme, Nexviazyme, Nexviadyme
  Groups: Other Enyzme Replacement Therapy (ERT)-treated patients
Other: Untreated — Patients who are not currently receiving any medical therapy for Pompe disease.
  Groups: Untreated patients (those who are not currently receiving any medical therapy for Pompe disease)

SUMMARY:
This is a global, multicenter, prospective, observational registry of patients with Pompe disease, including those with late-onset pompe disease (LOPD) and infantile-onset pompe disease (IOPD). Both untreated patients and those being treated with an approved therapy for Pompe disease are eligible to participate.

The objectives of the registry are:

* To evaluate the long-term safety of Pompe disease treatments through collection of data that describe the frequency of adverse events (AEs)/serious adverse events (SAEs) occurring in Pompe disease patients
* To evaluate the long-term real-world effectiveness of Pompe disease treatments
* To evaluate the long-term real-world impact of Pompe disease treatments on quality of life (QOL) and patient-reported outcomes (PROs)
* To describe the natural history of untreated Pompe disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LOPD or IOPD based on documented deficiency of GAA enzyme activity and/or GAA genotyping

Exclusion Criteria:

* Patients who are currently receiving investigational therapy for Pompe disease in a clinical trial, a compassionate use program, or an expanded access program (EAP)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population in this registry will consist of patients with a diagnosis of Pompe disease (LOPD or IOPD) based on documented deficiency of acid α-glucosidase (GAA) enzyme activity and/or GAA genotyping, regardless of time since diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2034-12-20 (Estimated); Study Completion 2034-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate long-term safety of Pompe disease treatments | 5 years
  Data collection that describe the frequency of AEs/SAEs occurring in Pompe disease patients

CONTACTS AND LOCATIONS:
Locations (41):
- United States (15):
  - University of Arkansas Medical Science, Little Rock, Arkansas
  - University of California Irvine, Irvine, California
  - Wolfson Children's Hospital, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, IU Health Physicians Neurology, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Neurogenetics, NYU Langone Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc., Fairfax, Virginia
- Medizinische Universitaet Wien, Vienna, Austria
- Laboratory for Muscle Diseases and Neuropathies, Leuven, Belgium
- Aarhus Universitets hospital, Aarhus C, Denmark
- Germany (5):
  - Ruhr-Universität Bochum im St. Josef-Hospital, Bochum
  - SphinCS, Institute of Clinical Science in LSD, Höchheim
  - Universitätsklinikum Gießen und Marburg GmhH, Marburg
  - Universitat Munchen - Friedrich Baur Institut, München
  - Universitaetsklinikum Ulm, Ulm
- Eginition Hospital, Athens, Greece
- Hungary (2):
  - University of Pécs, Pécs
  - University of Szeged, Szent-Györgyi Albert Clinical Center, Szeged
- Italy (4):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Centre of Expertise for muscular diseases and peripheral neuropathies European Reference Network for Rare Neuromuscular Diseases, Napoli
  - Department of Neurosciences Rita Levi Montalcini, University of Torino, Torino
  - Regional Coordinating Centre for Rare Diseases, university Hospital of Udine, Udine, Italy, Udine
- Dept of Pediatrics Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- entrum Medyczne Medyk, Rzeszów, Poland
- University Medical Centre Ljubljana, Institute of Clinical Neurophysiology, Ljubljana, Slovenia
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Cambridge University - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff, Cardiff
  - University Hospital of Wales, Cardiff
  - National Hospital for Neurology and Neurosurgery, London
  - Great Ormond Street Hospital NHS Foundation Trust, London
  - Royal Free Hospital NHS Foundation Trust, Manchester
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No